CLINICAL TRIAL: NCT02091206
Title: A Double Blind, Placebo-controlled, Two-part Study to Investigate the Dose-ranging Safety and Pharmacokinetics, Followed by the Efficacy and Safety of Cannabidiol (GWP42003-P) in Children and Young Adults With Dravet Syndrome
Brief Title: A Dose-ranging Pharmacokinetics and Safety Study of GWP42003-P in Children With Dravet Syndrome (GWPCARE1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1332 Part A; 2014-002941-23 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Dravet Syndrome
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GWP42003-P 5 mg/kg/day Dose (Experimental): Participants received GWP42003-P 5 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 5 mg/kg/day over 3 days and remained at this dose for the rest of the 21-day treatment period (19 days). The 21-day treatment period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P 5 mg/kg/day Dose
- GWP42003-P 10 mg/kg/day Dose (Experimental): Participants received GWP42003-P 10 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 10 mg/kg/day over 7 days and remained at this dose for the rest of the 21-day treatment period (15 days). The 21-day treatment period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P 10 mg/kg/day Dose
- GWP42003-P 20 mg/kg/day Dose (Experimental): Participants received GWP42003-P 20 mg/kg/day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 20 mg/kg/day over 11 days and remained at this dose for the rest of the 21-day treatment period (11 days). The 21-day treatment period was followed by a 10-day taper (10% per day) period.
  Interventions: Drug: GWP42003-P 20 mg/kg/day Dose
- Placebo (Placebo Comparator): Participants received placebo (0 mg/mL CBD), volume matched to one of the 3 dose levels (5, 10, or 20 mg/kg/day), administered orally, half in the morning and half in the evening for 21 days. To maintain the blinded aspect of the study, participants titrated the placebo dose over 3 to 11 days according to the matched investigational medicinal product (IMP) group (3, 7, and 11 days for the 5, 10, or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the rest of the 21-day treatment period. The 21-day treatment period was followed by a 10-day taper (10% per day of the matched dose) period.
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: GWP42003-P 5 mg/kg/day Dose — GWP42003-P was an oral solution containing 25 mg/milliliter (mL) cannabidiol (CBD) or 100 mg/mL CBD dissolved in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL). Participants were randomly assigned to receive either 5, 10 or 20 mg/kg/day.
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 5 mg/kg/day Dose
Drug: Placebo control — Placebo oral solution contained the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: Placebo
  Arms: Placebo
Drug: GWP42003-P 10 mg/kg/day Dose — GWP42003-P was an oral solution containing 25 mg/mL CBD or 100 mg/mL CBD dissolved in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL). Participants were randomly assigned to receive either 5, 10 or 20 mg/kg/day.
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 10 mg/kg/day Dose
Drug: GWP42003-P 20 mg/kg/day Dose — GWP42003-P was an oral solution containing 25 mg/mL CBD or 100 mg/mL CBD dissolved in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL). Participants were randomly assigned to receive either 5, 10 or 20 mg/kg/day.
  Other Names: Cannabidiol; Epidiolex
  Arms: GWP42003-P 20 mg/kg/day Dose

SUMMARY:
To evaluate the safety and pharmacokinetics (PK) of multiple doses of GWP42003-P compared with placebo in children with Dravet syndrome.

DETAILED DESCRIPTION:
This multi-center study consisted of 2 parts: Part A and Part B. Only Part A is described in this record. Part A was a randomized, double-blind 21-day treatment study period. Participants were randomized to one of 3 doses of active drug or placebo at a 4:1 ratio.

Participants who satisfied all inclusion and none of the exclusion criteria were assigned a unique participant number and then began a 28-day baseline observation period.

Eligible participants were then randomly assigned to receive one of 3 dose levels of GWP42003-P: 5 milligrams (mg) per kilogram (kg) per day, 10 mg/kg/day, 20 mg/kg/day, or matching placebo.

There were three groups of ten participants. In each group, participants were randomly assigned so that eight participants received active treatment and two participants received placebo. Participants received GWP42003-P or placebo for a 21-day exposure period, which consisted of a titration period, followed by a stable dose period.

A PK assessment took place after the first single dose of GWP42003-P. There was a second PK assessment after 21 days of consecutive dosing with GWP42003-P. Participants who took clobazam (CLB) as an adjunctive treatment were asked to take their usual dose 2 hours prior to attending the clinic. The same recommendation was made for other concomitant antiepileptic drugs (AEDs), if applicable. This was so that the pre-treatment (with GWP42003-P) plasma concentrations of CLB, its major metabolite N-desmethylclobazam, and any other concomitant AEDs could be measured, and the impact of GWP42003-P treatment on these levels evaluated. Interim clinic visits to (primarily) evaluate safety and adherence to the titration regimen took place at 7 and 14 days of treatment.

After 21 days of treatment, all participants commenced a 10-day down-titration taper period. An independent Data Safety Monitoring Committee reviewed unblinded safety and PK data and recommended the target dose (up to 20 mg/kg/day) for Part B of the study and for an open label extension study. Once the safety review of Part A data had taken place, participants had the option of entering the open label extension study.

A follow-up telephone call was made 28 days after the end of dosing for participants who did not enter the open label extension study within this time-frame.

Throughout the 21-day treatment period and the 10-day taper period, there were regular safety telephone calls (approximately every 2 days) to check participant status. Weekly safety telephone calls were made during the 28-day follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants were male or female aged between 4 and 10 years (inclusive).
* Participants had a documented history of Dravet Syndrome that was not completely controlled by AEDs.
* Participants took one or more AEDs at a dose which had been stable for at least 4 weeks.
* Participants had experienced fewer than 4 convulsive seizures (tonic-clonic, tonic, clonic, atonic seizures) during the 28-day baseline period.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation [VNS]) were stable for four weeks prior to screening and participants were willing to maintain a stable regimen throughout the study. The ketogenic diet and VNS treatments were not counted as an AED.

Key Exclusion Criteria:

* Participants had clinically significant unstable medical conditions other than epilepsy.
* Participants had clinically relevant abnormalities in the 12-lead electrocardiogram measured at screening or randomization.
* Participants were currently using or had in the past used recreational or medicinal cannabis, or synthetic CBD based medications (including Sativex®) within the 3 months prior to study entry and were unwilling to abstain for the duration for the study.
* Participants had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP.
* Participants who had been part of a clinical trial involving another investigational product in the previous 6 months.
* There were plans for the participants to travel outside their country of residence during the study.
* Participants were previously randomized into this study. In particular, participants participating in Part A of the study cannot enter Part B.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2015-03-09 (Actual); Study Completion 2015-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Houston, Texas
- United Kingdom (3):
  - Edinburgh
  - Liverpool
  - London

REFERENCES:
- [Background] Devinsky O, Patel AD, Thiele EA, Wong MH, Appleton R, Harden CL, Greenwood S, Morrison G, Sommerville K; GWPCARE1 Part A Study Group. Randomized, dose-ranging safety trial of cannabidiol in Dravet syndrome. Neurology. 2018 Apr 3;90(14):e1204-e1211. doi: 10.1212/WNL.0000000000005254. Epub 2018 Mar 14. PMID 29540584

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003-P 5 mg/kg/Day Dose: Participants received GWP42003-P 5 milligrams (mg) per kilogram (kg) per day administered orally, half in the morning and half in the evening. Participants titrated GWP42003-P to 5 mg/kg/day over 3 days and remained at this dose for the rest of the 21-day treatment period (19 days). The 21-day treatment period was followed by a 10-day taper (10% per day) period.
- Placebo: Participants received placebo (0 mg/milliliter [mL] cannabidiol [CBD]), volume matched to one of the 3 dose levels (5, 10, or 20 mg/kg/day), administered orally, half in the morning and half in the evening for 21 days. To maintain the blinded aspect of the study, participants titrated the placebo dose over 3 to 11 days according to the matched investigational medicinal product (IMP) group (3, 7, and 11 days for the 5, 10, or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the rest of the 21-day treatment period. The 21-day treatment period was followed by a 10-day taper (10% per day of the matched dose) period.
Period: Treatment Period
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo
Started | 10 | 8 | 9 | 7
Safety Analysis Set (All randomized participants who received at least 1 dose of IMP) | 10 | 8 | 9 | 7
Completed | 10 | 7 | 8 | 7
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Met withdrawal criteria | 0 | 0 | 1 | 0
Period: Taper Period
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo
Started | 10 | 7 | 8 | 7
Completed | 9 | 7 | 8 | 5
Not Completed | 1 | 0 | 0 | 2
Not completed — Participant refused study drug | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: included all participants randomized to treatment who received at least 1 dose of IMP. Participants were analyzed according to the treatment they received. Only participants for whom it had been confirmed that they did not take any IMP were excluded from the safety analysis set.
Groups:
- Placebo: Participants received placebo (0 mg/mL CBD), volume matched to one of the 3 dose levels (5, 10, or 20 mg/kg/day), administered orally, half in the morning and half in the evening for 21 days. To maintain the blinded aspect of the study, participants titrated the placebo dose over 3 to 11 days according to the matched IMP group (3, 7, and 11 days for the 5, 10, or 20 mg/kg/day GWP42003-P groups, respectively) and remained at this dose for the rest of the 21-day treatment period. The 21-day treatment period was followed by a 10-day taper (10% per day of the matched dose) period.
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo | Total
Number analyzed (Participants) | 10 | 8 | 9 | 7 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.150 (1.8955) | 7.368 (2.1229) | 8.671 (1.7957) | 6.978 (0.9476) | 7.568 (1.8300)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 2 | 18
  Male | 5 | 3 | 3 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) with an onset date on or after the first dose of IMP. If an AE had a partial onset date and it was unclear from the partial date (or the stop date) whether the AE started prior to or following the first dose of IMP then the AE was considered a TEAE. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through the Safety Follow-up Visit (Day 60) is presented.
  A summary of serious and all other non-serious AEs regardless of causality is located in the Adverse Events module.
Time Frame: Baseline (Day 1) through Safety follow-up visit (Day 60)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 8 | 9 | 7
Participants | 2 | 1 | 0 | 1

2. Secondary Outcome: Area Under The Concentration-Time Curve Calculated To The Last Observable Concentration At Time T (AUC0-t) For CBD And Its Metabolites At Days 1 And 22
Description: AUC0-t for CBD and its major metabolites, 6-hydroxy-CBD (6-OH-CBD), 7-hydroxy-CBD (7-OH-CBD), and 7-carboxy-CBD (7-COOH-CBD) were calculated using blood samples collected before and after IMP dosing on Days 1 and 22. One sample was collected predose, 2 to 3 hours postdose, and 4 to 6 hours postdose for CBD and its metabolites. Results are presented for participants who received GWP42003-P at 5, 10, or 20 mg/kg/day during the study and for participants with a numeric result for the given evaluation.
Time Frame: Predose and 2-6 hours postdose on Days 1 and 22
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanograms/mL
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose
Number analyzed (Participants) | 10 | 8 | 9
hours * nanograms/mL
  Day 1 CBD: number analyzed (Participants) | 5 | 7 | 7
  Day 1 CBD | 70.61 (20.38) | 66.35 (120.8) | 73.69 (96.64)
  Day 22 CBD: number analyzed (Participants) | 9 | 7 | 7
  Day 22 CBD | 240.8 (100.8) | 721.8 (79.92) | 962.6 (93.43)
  Day 1 6-OH-CBD: number analyzed (Participants) | 3 | 5 | 5
  Day 1 6-OH-CBD | 3.27 (132) | 2.79 (87.7) | 5.16 (57.2)
  Day 22 6-OH-CBD: number analyzed (Participants) | 8 | 7 | 6
  Day 22 6-OH-CBD | 9.33 (119) | 26.3 (82.9) | 58.6 (90.1)
  Day 1 7-OH-CBD: number analyzed (Participants) | 5 | 7 | 8
  Day 1 7-OH-CBD | 21.9 (57.0) | 18.4 (299) | 30.2 (105)
  Day 22 7-OH-CBD: number analyzed (Participants) | 8 | 7 | 6
  Day 22 7-OH-CBD | 131 (107) | 244 (120) | 508 (96.0)
  Day 1 7-COOH-CBD: number analyzed (Participants) | 6 | 6 | 6
  Day 1 7-COOH-CBD | 297 (97.3) | 125 (1750) | 195 (573)
  Day 22 7-COOH-CBD: number analyzed (Participants) | 9 | 5 | 5
  Day 22 7-COOH-CBD | 4190 (81.20) | 9220 (178) | 15500 (148)

3. Secondary Outcome: Mean Percentage Change From Baseline To End Of Treatment In Plasma Clobazam (CLB) And N-Desmethylclobazam (N-CLB) Concentrations
Description: Plasma concentrations of CLB and N-CLB were measured on Days 1 and 22. Participants were instructed to take their daily dose of CLB 2 hours prior to the anticipated pre-IMP blood specimen collection on both days. Blood samples were collected prior to administration of IMP. Results are presented for a subgroup of participants who took CLB during the study and had PK samples analyzed at both PK sampling visits (Days 1 and 22).
Time Frame: Predose on Days 1 and 22
Population: as for baseline characteristics
Measure: Number; unit: percent change
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5
percent change
  % change in CLB | -1.2 | 18.0 | 29.6 | 15.1
  % change in N-CLB | 258.7 | 170.7 | 228.9 | -5.6

ADVERSE EVENTS:
Time Frame: Up to Day 60
Description: All participants randomized to treatment who received at least 1 dose of IMP. Participants were analyzed according to the treatment they received. Only participants for whom it had been confirmed that they did not take any IMP were excluded from the safety analysis set.
Arm/Group | GWP42003-P 5 mg/kg/Day Dose | GWP42003-P 10 mg/kg/Day Dose | GWP42003-P 20 mg/kg/Day Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/8 | 1/9 | 1/7
Other Adverse Events (participants affected / at risk) | 8/10 | 5/8 | 7/9 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 5 mg/kg/Day Dose (N=10) | GWP42003-P 10 mg/kg/Day Dose (N=8) | GWP42003-P 20 mg/kg/Day Dose (N=9) | Placebo (N=7)
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Parvovirus Infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 5 mg/kg/Day Dose (N=10) | GWP42003-P 10 mg/kg/Day Dose (N=8) | GWP42003-P 20 mg/kg/Day Dose (N=9) | Placebo (N=7)
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Urine ketone body absent (Investigations) | 1 | 0 | 0 | 0
Urine ketone body present (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 1
Sedation (Nervous system disorders) | 2 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 2 | 3 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 3 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Analytical issues for 7-OH-CBD related to reference material batch used during analysis. Data are qualitative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days